CLINICAL TRIAL: NCT00248053
Title: Use of Curcumin in the Lower Gastrointestinal Tract in Familial Adenomatous Polyposis (FAP) Patients
Brief Title: Use of Curcumin in the Lower Gastrointestinal Tract in Familial Adenomatous Polyposis Patients
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Subsequent data generated by our collaborators have shown efficacy with curcumin and quercetin in 5 patients in a non placebo controlled trial.
Sponsor: Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Francis M. Giardiello, Professor of Medicine, Johns Hopkins University
Allocation: Non-Randomized | Model: Crossover | Masking: None
Other Study IDs: 05-04-12-04
Record Dates: First submitted 2005-11-01; First posted 2005-11-03 (Estimated); Last update posted 2012-09-20 (Estimated); Status verified 2012-09

CONDITIONS: Familial Adenomatous Polyposis
Keywords: Familial adenomatous polyposis patient with 5 or more adenomatous polyps in the colon or ileoanal pouch
MeSH Terms: conditions — Adenomatous Polyposis Coli | interventions — Curcumin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Lower GI (Other)
  Interventions: Drug: curcumin

INTERVENTIONS:
Drug: curcumin — curcumin 500 mg by mouth, three times a day for 9 months

SUMMARY:
The purpose of this study is to assess if curcumin, a commonly used food spice, can regress colorectal adenomatous polyps in patients with familial adenomatous polyposis, an inherited form of colorectal cancer.

ELIGIBILITY:
Inclusion Criteria:

* Familial adenomatous polyposis
* 18 years of age or older
* 5 or more adenomas of colorectum or ileum

Exclusion Criteria:

* Female patient of child bearing age not on effective birth control pills
* Pregnant women
* White blood cell (WBC) count less than 4000
* Platelets (Plts) less than 100,000
* Blood urea nitrogen (BUN) greater than 25
* Creatine greater than 1.5
* Patients unable to stop non-steroidal anti-inflammatory drugs (NSAIDs) during duration of trial
* Malignancy
* Patient with active bacterial infections of gastroesophageal reflux disease or peptic ulcer disease
* Patient on warfarin or anti-platelet drugs

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2005-11; Primary Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
polyp number and size | one year

SECONDARY OUTCOMES:
side effects and medication compliance | one year

CONTACTS AND LOCATIONS:
Overall Officials: Francis M Giardiello, M.D., Principal Investigator — Johns Hopkins University